CLINICAL TRIAL: NCT05929820
Title: Pilot Randomized Controlled Trial Assessing the Impact of Protect Your Colon™ on Colorectal Cancer Screening Behaviors
Brief Title: Impact of Protect Your Colon™ on CRC Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Almario, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STUDY2402
Record Dates: First submitted 2023-05-18; First posted 2023-07-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Screening
Keywords: Decision aid; Stool test; Colonoscopy; CT scan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protect Your Colon™ (Intervention) (Experimental): Patients randomized to Protect Your Colon™ will be directed to go through the website before their clinic appointment. Those who finish the decision aid will then review their personalized report which details their priorities in selecting a screening test as well as the test that best matches their values. Patients will also be encouraged to bring their personalized report with them to the visit to discuss with their doctor. All intervention participants will also receive a reminder via email one day before their scheduled clinic visit. They will be reminded to go through the Protect Your Colon™ website before the clinic visit and to bring their personalized report with them to the visit.
  Interventions: Behavioral: Protect Your Colon™
- Usual Care (Control) (No Intervention): The usual care group will be managed according to the providers' customary practices: CRC screening discussions, if any, are at the discretion of the provider as Cedars-Sinai does not employ a standardized approach. Patients randomized to the control arm will not be sent any materials before their clinic appointment.

INTERVENTIONS:
Behavioral: Protect Your Colon™ — Protect Your Colon™ is an online decision aid focused on CRC screening. The site will first educate patients on the importance of CRC screening and offer information on the advantages and disadvantages of the available test options. Protect Your Colon™ will then present an interactive conjoint analysis-a quantitative survey technique that elucidates how individuals make complex decisions-to precisely determine individuals' latent preferences regarding CRC screening options. Afterwards, the app will generate a personalized report that rank orders the importance of each test attribute (e.g., accuracy, invasiveness, test frequency) in patients' decision making and identifies the screening modality that best matches their preferences. The report will also be shareable with physicians, enabling patients and providers to engage in shared decision making surrounding CRC screening in the clinic.
  Arms: Protect Your Colon™ (Intervention)

SUMMARY:
The purpose of the research is to assess the impact of Protect Your Colon™, a colorectal cancer (CRC) screening decision aid, on patients' CRC screening behaviors. The Investigators hypothesize that Protect Your Colon™, through optimizing shared decision making, will lead to selection of a test that accurately matches patients' values and increase CRC screening uptake. To test this hypothesis, the investigators will conduct a pilot randomized controlled trial (RCT) to assess if provision of Protect Your Colon™ improves communication on CRC screening, intent to complete screening, and ultimately uptake of screening vs. usual care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 45 to 75 years old
* No prior CRC screening or not up-to-date with CRC screening
* Not at high risk for CRC (e.g., inflammatory bowel disease, colon polyposis syndromes, family history of CRC)
* No prior colon polyps
* Additional inclusion criteria for participants recruited through Cint online survey panels: (i) appointment with a primary care provider up to 6 weeks from time of screening, and (ii) have Preferred Provider Organization (PPO) insurance.

Exclusion Criteria:

* Does not speak English
* Does not have internet access
* Any records flagged "break the glass" or "research opt out."

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of completion of a CRC screening test | 6 months post visit
  Uptake of CRC screening within 6 months of patients' initial visit

SECONDARY OUTCOMES:
Qualitative feedback on details of CRC screening test | 1 day post visit
  Completion of questionnaire that looks at:
  * Whether CRC screening discussions took place during the visit
  * What specific CRC screening tests were discussed during the visit
  * Patient's intent to complete CRC screening
  * Patient's perceptions on feeling informed about the alternatives, benefits, and risks of the different screening options as well as their clarity on their personal values
  * Patient's assessment of shared decision making on CRC screening
  * Intervention patients' assessment of the usefulness of Protect Your Colon™

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Almario, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigator (Christopher V. Almario) upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after study completion and for up to 3 years after study completion.
Access Criteria: The data that support the findings of this study will be available from the principal investigator (Christopher V. Almario) upon reasonable request.